CLINICAL TRIAL: NCT01997021
Title: Effects of Interrupting Sedentary Time on Glycemic Control in Older Overweight and Obese Adults
Acronym: B-WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-2594
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Syndrome; Diabetes; Aging
Keywords: Sedentary behavior; physical activity; older adults
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- US/IW/CW (Experimental): This is a 3 arm crossover design. Arm US/IW/CW corresponds to the group of participants randomized to uninterrupted sitting (US) first, then Intermittent Walking (IW) and then continuous walk (CW).
  Interventions: Other: US; Other: IW; Other: CW
- IW/US/CW (Experimental): This is a 3 arm crossover design. Arm IW/US/CW corresponds to the group of participants randomized to Intermittent Walking (IW) first, then uninterrupted sitting (US), and then continuous walk (CW).
  Interventions: Other: US; Other: IW; Other: CW
- IW/CW/US (Experimental): This is a 3 arm crossover design. Arm IW/CW/US corresponds to the group of participants randomized to Intermittent Walking (IW) first, then Continuous Walk (CW) and then Uninterrupted Sitting (US).
  Interventions: Other: US; Other: IW; Other: CW
- CW/IW/US (Experimental): This is a 3 arm crossover design. Arm CW/IW/US corresponds to the group of participants randomized to Continuous Walk (CW) first, then Intermittent Walking (IW) and then Uninterrupted Sitting (US).
  Interventions: Other: US; Other: IW; Other: CW
- CW/US/IW (Experimental): This is a 3 arm crossover design. Arm CW/IW/US corresponds to the group of participants randomized to Continuous Walk (CW) first, then Uninterrupted Sitting (US), and then Intermittent Walking (IW).
  Interventions: Other: US; Other: IW; Other: CW
- US/CW/IW (Experimental): This is a 3 arm crossover design. Arm US/CW/IW corresponds to the group of participants randomized to Uninterrupted Sitting (US) first, then Continuous Walk (CW), and then Intermittent Walking (IW).
  Interventions: Other: US; Other: IW; Other: CW

INTERVENTIONS:
Other: US — US is a 5-hour intervention/condition where participants will be required to sit quietly for 5 consecutive hours.
  Other Names: Uninterrupted sitting
Other: IW — IW is a 24-hour intervention/condition where participants interrupt sedentary time with short 1.5 minute walking bout.
  Other Names: Intermittent Walking
Other: CW — CW is a 24-hour intervention/condition where participants perform a 36 minute continuous walking bout and are seated the remainder of the time.
  Other Names: Continuous Walking

SUMMARY:
Increasing physical activity in older adults has important implications for treating obesity related metabolic conditions, however the interaction of aging- and obesity-related declines in physical function may make adding structured exercise particularly challenging for this group. Given these challenges, an alternative prescription to traditional structured exercise, may be short bouts of intermittent walking scattered throughout the day - this may be an effective strategy to increase physical activity, reduce sedentary behavior, and improve glycemic control in overweight/obese older adults. The purpose of this project is to determine how interrupting sedentary time with short bouts of moderate intensity walking affects important metabolic outcomes in older, overweight adults. It would also be of interest to compare the effects of short, frequent interruptions in sedentary behavior to a traditional exercise prescription (continuous 30 min walking bout) on metabolic outcomes (e.g., glycemic control, insulin sensitivity, and 24 h fat oxidation). Thus, the overall aims of the proposed research are to 1) Determine the effect of performing short bouts of moderate-intensity intermittent walking (IW) on glucose and insulin metabolism compared to uninterrupted sitting (US) in older overweight and obese adults. 2) To compare the effects of interrupting sedentary time (IW) vs. a traditional exercise prescription (continuous 30 m walk (CW)) on metabolism.

The investigators hypothesize that interrupting sedentary time with intermittent walking will improve glucose and insulin metabolism compared to uninterrupted sitting and it will be as effective at improving metabolism as a single continuous 30 min walk.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-85 yr • BMI 25-35 kg.m-2
* Non-exercisers (<150 m/wk of moderate intensity exercise)
* Sedentary (>60% of waking day sedentary)
* Able to walk on a treadmill for 36 continuous minutes at a pace of at least 2.0 mph

Exclusion Criteria:

* Self-reported acute or chronic disease (e.g. diabetes, heart disease, thyroid disease)
* Fasting plasma glucose ≥ 126 mg/dl - participants will not be excluded if they an abnormal post prandial glucose levels (e.g. glucose ≥ 200 mg/dl) following the MTT's.
* Tobacco use (cigarettes, cigars, or chewing tobacco) within the past 6 months
* Females who previously used (> 6 months) or are currently using any formulation of estrogen-based hormone therapy (e.g., oral Premarin, transdermal 17-estradiol, selective estrogen receptor modulators).
* Resting diastolic blood pressure > 100 mm mercury or resting systolic blood pressure > 160 mm mercury
* Contra-indications to exercise (e.g. orthopedic limitations)
* Unable to walk on a treadmill for 36 continuous minutes at a pace of at least 2.0 mph

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Incremental area under the glucose curve in response to meal tolerance test (MTT) | Hourly for 5 hours after meal is consumed
  Meal tolerance test is performed during uninterrupted sitting condition and during intermittent walking condition. Glucose area under the curve (AUC) is compared between conditions.
Area under the insulin curve in response to meal tolerance test | Hourly for 5 hours after meal is consumed
  Meal tolerance test is performed during uninterrupted sitting condition and during intermittent walking condition. Insulin AUC is compared between conditions.

SECONDARY OUTCOMES:
Postprandial glycemia in response to meal tolerance test | Continuously for 5 hours after meal is consumed
  Postprandial glycemia (PPG) will be measured using a continuous glucose monitor. Peak PPG, rate of change in peak PPG and duration of hyperglycemia will be calculated. Meal tolerance test will be performed during uninterrupted sitting condition and during intermittent walking condition. PPG will be compared between conditions.
Insulin sensitivity | Immediately post 24 hr intermittent walking and continuous walking conditions
  Insulin sensitivity will be measured using a hyperinsulinemic euglycemic clamp. IS will be assessed after intermittent walking condition and after continuous walk condition. IS will be compared between conditions.
24-hr Fat Oxidation | Continuously during 24 hr intermittent walking and continuous walking conditions
  Fat oxidation will be measured in a whole room indirect calorimeter during the intermittent walking condition and during the continuous walk condition. Fat oxidation will be compared between conditions.
24-hour Glycemic variability | Continuously during 24 hr intermittent walking and continuous walking conditions
  Glycemic variability will be measured using a continuous glucose monitor during the intermittent walking condition and during the continuous walk condition. Glycemic variability will be compared between conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lyden, PhD, Principal Investigator — University of Colorado, Denver; Ed Melanson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States